CLINICAL TRIAL: NCT04223453
Title: Body Composition in Patients With Acute Pneumonia Measured by Bioimpedance and DXA
Brief Title: Body Composition Measurements in Pneumonia
Status: Completed | Type: Observational
Sponsor: Jens Rikardt Andersen (Other)
Collaborators: Hillerod Hospital, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Other Study IDs: Daniel1
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Acute Infection Respiratory
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: BIA and DXA — Patients with acute pneumonia measured simultaneously with DXA-scan and BIA-impedance

SUMMARY:
The purpose of this study is to validate and standardize bioelectrical impedance analysis (BIA, Maltron BioScan touch i8) for estimating body composition in hospitalized elderly patients with pneumonia. Body composition assessments with BIA and dual-energy x-ray absorptiometry (DXA,

DETAILED DESCRIPTION:
Holigic Discovery) was performed on 36 non-fasting patients over 65 years of age. 29 patients had BIA performed within 24 hours after hospital admission and at the date of discharge. 17 patients had BIA performed in fasted state and one hour after an intake of 300 ml glucose solution.

ELIGIBILITY:
Inclusion Criteria:

* Acute pneumonia,
* Accept participation (informed consent)
* Understand the given instructions and information

Exclusion Criteria:

* None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: X-ray verified acute pneumonia > 65 years of age
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between LBM (lean body mass) with DXA and BIA | within 3 days
  At admittance both methods.

SECONDARY OUTCOMES:
Development in lean-body-mass during hospital stay | 3-10 days (hospital stay)
  Repeated measurement with BIA during the state of acute infection
BIA measured before and after oral glucose load test | 1 hour
  To investigate for the effect of fasting on the determination of total body water with BIA

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Principal Investigator — University of Copenhagen, Department of Nutrition, Exercise and Sports
Locations (1):
- Hillerød Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No